CLINICAL TRIAL: NCT00120120
Title: A Multicenter, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Lenalidomide in the Treatment of Painful Lumbar Radiculopathy
Brief Title: Study to Evaluate the Efficacy and Safety of Lenalidomide in the Treatment of Painful Lumbar Radiculopathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Victor Sloan MD, VP Clinical R&D, Rheumatology, Celgene Corporation
Organization: Celgene (Industry)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-5013-RAD-001
Record Dates: First submitted 2005-07-08; First posted 2005-07-15 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Radiculopathy
Keywords: Radiculopathy; Back Pain; Lumbar Pain; CC-5013; Revlimid; Lenalidomide
MeSH Terms: conditions — Radiculopathy; Back Pain; Low Back Pain | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Lenalidomide (CC-5013)
- 2 (Experimental)
  Interventions: Drug: Lenalidomide (CC-5013)

INTERVENTIONS:
Drug: Lenalidomide (CC-5013) — Lenalidomide 2-5 mg capsules taken one time per day
  Other Names: Revlimid

SUMMARY:
The purpose of this multicenter, double-blind, placebo-controlled study is to evaluate the efficacy and safety of lenalidomide in the treatment of painful lumbar radiculopathy.

DETAILED DESCRIPTION:
Study Duration: Pre-randomization Phase: 14 days; Treatment Phase: 12 weeks; Extension Phase: Ongoing; Total Study Duration: Up to 14 weeks + the duration of the extension phase

For each subject, the study consists of three phases: Pre-randomization phase (14 days), Treatment Phase (12 weeks) and an extension phase where subjects have the opportunity to receive lenalidomide treatment as long as benefit is derived from the drug. Subjects who complete all 12 weeks of the treatment phase may be eligible to initiate (subjects randomized to receive placebo in the treatment phase) or continue to receive lenalidomide therapy (subjects randomized to receive lenalidomide in the treatment phase) in the extension phase. Subjects may continue in the extension phase as long as a benefit is derived from the drug.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater at the time of signing the informed consent form
* Clinical diagnosis of painful radiculopathy which is based on the presence of pain in the distribution of the sciatic nerve or L4, L5 or S1 dermatomes. The pain must be primarily in the lower leg and radiate to the ankle or foot.
* History of painful radiculopathy involving one or both of the distal lower extremities for greater than or equal to 6 months
* MRI or CT scan within the past 2 years or more recent if symptoms have changed
* Positive straight leg raising (SLR) test in the index ipsilateral leg (pain radiating below the knee at an elevation of <60 degrees). In the presence of bilateral leg pain, the leg with the most severe pain will be designated the index leg.
* Screening (Visit 1): Radiculopathy PI-NRS score must be at least 5 on an 11-point (0-10) PI-NRS
* Randomization (Visit 2): Average radiculopathy PI-NRS score for randomization purposes will be based on AM and PM assessments made during the 7 days prior to randomization:

  1. At least eight radiculopathy PI-NRS scores during this 7-day period are required and
  2. Average radiculopathy PI-NRS score during this period must be at least 5 on an 11-point (0-10) PI-NRS.
* Stable doses of tricyclic antidepressants, AEDs, mexiletine hydrochloride, dextromethorphan, capsaicin, NSAIDs, opioids or other medications (including prn radiculopathy medication usage) that could affect symptoms of painful radiculopathy for at least 28 days prior to randomization (Visit 2).
* Negative drugs of abuse screen (except drugs known to be prescribed for radiculopathy).
* Women of childbearing potential (WCBP) must agree to practice complete abstinence from heterosexual intercourse or to use two methods of contraception beginning 4 weeks prior to the start of study drug (Day 1) while on study drug (including dose interruptions) and 4 weeks after the last dose of study drug. The two methods of contraception must include one highly effective method (i.e. intrauterine device, hormonal [birth control pills, injections, or implants only if used in conjunction with a low-dose (81 mg/day) aspirin regimen], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e. latex condom, diaphragm, cervical cap). If a hormonal method (birth control pills, injections or implants) or IUD is not medically possible for the subject, two of the barrier methods will be acceptable.
* Women of childbearing potential (WCBP) must have two negative pregnancy tests (sensitivity of at least 50 mlU/mL) prior to starting study drug treatment. The first test should be performed within 10-14 days and the second within 24 hours of starting study drug. Once treatment has started, it is recommended that subjects have weekly pregnancy tests during the first 4 weeks of treatment. Thereafter, subjects are required to have pregnancy testing every 4 weeks in females with regular menstrual cycles and every 2 weeks in females with irregular cycles.
* Males (including those who have had a vasectomy) must use barrier contraception (latex condoms) when engaging in reproductive sexual activity with WCBP while on study drug and for 4 weeks after the last dose of study drug.

Exclusion Criteria:

* Pain localized in the low back or other sites that is a greater component of subject's total pain problem than lower leg and foot pain
* Ankle or foot problems, which could interfere with the assessment of radiculopathy pain
* Unstable lumbar spinal segment
* Evidence of an acute operable lesion or tumor based on CT-scan or MRI results
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac or neurological disease
* Any medical condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Presence of a clinically significant psychiatric diagnosis(es) that would impair reliable study participation
* History of deep vein thrombosis (DVT) or stroke in the past 5 years
* History of low back or lumbar spinal surgery
* Documented metabolic or toxic peripheral neuropathies
* Any other serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from understanding or signing the informed consent form
* White blood cell count (WBC) < 3.5 x 10/L at Visit 1
* Bilirubin, alanine transaminase (ALT), aspartate transaminase (AST) or alkaline phosphatase values more than two times the upper limit of the normal range at Visit 1
* Abnormal T3, T4 or TSH test value(s) at Visit 1 (An abnormal TSH level in the presence of normal T3 and T4 levels is acceptable).
* More than 6 epidural steroid injections within the 12 months prior to randomization (Visit 2).
* Use of an epidural steroid injection within 28 days of randomization
* Concurrent use of a spinal cord stimulator or intrathecal drug infusion device
* Limited duration (planned termination during either the Pre-randomization or Treatment Phases) non-drug therapies (including physical therapy, acupuncture and chiropractic treatments) during the Pre-randomization and Treatment Phases of the study. Subjects may continue to do home exercises, if they have been a stable part of the subject's treatment regimen for at least 28 days prior to randomization.
* Use of concomitant medications, which could increase the risk for developing DVT, except for steroid-based contraceptives (oral, injectable, implantable) and hormone replacement therapies only if used in conjunction with a low-dose (81 mg/day) aspirin regimen
* Use of oral corticosteroids (except for asthma inhalers and Medrol Dosepak) within 28 days prior to randomization
* Concurrent use of thalidomide
* Prior development of an allergic reaction/hypersensitivity, a moderate or severe rash, or any desquamation while taking thalidomide.
* Prior treatment with lenalidomide
* Use of any other experimental drug or therapy within 28 days of the start of the Treatment Phase
* Current pregnancy or lactation
* History of poor compliance or the inability to comply with medical regimens or study requirements
* Inability to use an electronic diary
* Active litigation (i.e. any pending litigation or pending proceeding), compensation or disability issues related to painful radiculopathy (Subjects whose cases have been settled or finally decided are eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2005-01; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in RAD pain intensity ratings using PI-NRS | baseline to week 12

SECONDARY OUTCOMES:
Safety (type, frequency, severity, and relationship to study drug) | change from baseline
Change from baseline in the PM PI NRS value | change from baseline
Change from baseline in the AM PI NRS value | change from baseline
Change from baseline inactivity level rating using an NRS | change from baseline
Change from baseline in SLR angle of elevation without induced pain | change from baseline
Change from baseline in the SF-MPQ total score and subscale scores | change from baseline
Changes from baseline in the BPI score relative to baseline pain ratings and interference scales | change from baseline
Changes from baseline in the POMS total mood score and six dimension subscale scores | change from baseline
Change from baseline in the PDI score | change from baseline
Change from baseline in the Modified Oswestry Low Back Pain Disability Questionnaire total score | change from baseline
Patient global impression of change | change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Victor Sloan, MD, Study Director — Celgene Corporation
Locations (23):
- United States (23):
  - Arizona Research Center, Phoenix, Arizona
  - Genova Clinical Research, Inc, Tucson, Arizona
  - Loma Linda Institution, Loma Linda, California
  - Space Coast Neurology, Palm Bay, Florida
  - Gold Coast Research, LLC, Weston, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Rehab Institute of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins Pain Center, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Pain Mgmt Ctr, St Louis, Missouri
  - North Shore University Hospital, Bethpage, New York
  - University of Rochester Medical CenterPain Services, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Carolinas Pain Institute, P.A. & the Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - Research Institute of Greater Dayton, Dayton, Ohio
  - Attn: Maryjane CerroneLehigh Valley Hospital, Allentown, Pennsylvania
  - Drexel University College of MedicineDepartment of Neurology Rm 7102, Philadelphia, Pennsylvania
  - Texas Tech Medical Center Department of Anesthesiology, Lubbock, Texas
  - KRK Medical Research, Richardson, Texas
  - Fletcher Allen Healthcare for Pain Medicine, South Burlington, Vermont
  - University of Virginia Pain Management Center, Charlottesville, Virginia
  - Swedish Pain Services, Seattle, Washington

REFERENCES:
- [Derived] Manning DC, Gimbel J, Wertz R, Rauck R, Cooper A, Zeldis JB, Levinsky DM. A Phase II Randomized, Double-Blind, Placebo-Controlled Safety and Efficacy Study of Lenalidomide in Lumbar Radicular Pain with a Long-Term Open-Label Extension Phase. Pain Med. 2017 Mar 1;18(3):477-487. doi: 10.1093/pm/pnw212. PMID 27550953